CLINICAL TRIAL: NCT04849923
Title: Validation of a Digital Twin to Predict the Adaptation of Muscle Strength and Muscle Size Due to Strength Training
Brief Title: Validation of a Digital Twin Performing Strength Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Swiss Federal Institute of Sport Magglingen (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Digital Twin
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Healthy
Keywords: strength training
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: controll group, two groups of strength training with different effort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- controll group (No Intervention): This group has no additional strength training
- 1 training per week (Experimental): This group performs one strength training session per week
  Interventions: Other: Strength training session
- 3 trainings per week (Experimental): This group performs two strength training sessions per week
  Interventions: Other: Strength training session

INTERVENTIONS:
Other: Strength training session — Conduct of an 8-week strength training intervention of key muscle-tendon groups associated with knee joint stability in the training-specific setting of each participant. Participants are randomly allocated into three study groups with increasing levels of loading (Group#1: no training, Group#2: 1 training per week, Group#3: 3 trainings per week) with the same number of subjects and gender distribution in each group (n=12 per group, 6F and 6M). The same guidelines for the warm-up and the type of exercises will be given prior to the intervention study to each participant. Participants are asked to record exercise load and volume as well as monitor training-related variables and 1RM using the iOS Strength Control app. Participants perform the strength training self-directedly in their chosen fitness/training facilities as it fits into their weekly routine. Contact to the study investigator is ensured at all times in case of questions.
  Other Names: resistance training
  Arms: 1 training per week; 3 trainings per week

SUMMARY:
Background: Muscular strength training interventions have long been a cornerstone in the prevention, non-surgical management and rehabilitation of the entire spectrum of musculoskeletal injuries and diseases. The key goal of strength training, especially during rehabilitation, is to regain healthy musculoskeletal function. Yet, there remains a fundamental lack of understanding with regards to the relationship between subject-specific musculoskeletal biomechanics (i.e. multi-body dynamics function) and different types of strength training interventions because of limitations in assessing these parameters outside the research setting. Thus, clinicians, physiotherapists and coaches continue making training recommendations based on subjective and generalised guidelines, with ineffective or possibly harmful consequences for individual patients and athletes.

Goal: This project aims to advance strength training guidelines and monitoring of training safety and efficiency by means of subject-specific anatomically-based modelling, biomechanical analysis of musculoskeletal function and mobile monitoring of training volume and muscular fatigue in the athletic and recreational setting.

Method: For validation purposes, the investigators will conduct an 8-week intervention study in healthy volunteers with three levels of strength training volume of the key muscle-tendon groups associated with knee joint stability and relate the changes in musculoskeletal and biomechanical parameters to the training-specific parameters and muscular fatigue from mobile monitoring through correlation analysis.

Relevance: In Switzerland, more than 1.3 Mio people are members of a fitness center. Strength training is not only a cornerstone in the maintenance of fitness and rehabilitation from musculoskeletal injuries and diseases as the most frequently reported health issues.

DETAILED DESCRIPTION:
Hypothesis: It is hypothesized that advanced subject-specific musculoskeletal modelling in combination with mobile monitoring technology as embedded in the iPhone and Apple Watch allow for accurate prediction of changes in muscle strength and muscle size in the lower limbs following an 8-week strength training intervention of key muscle-tendon groups associated with knee joint stability.

Primary Objective: Prediction of changes in muscle strength in the lower limbs due to different strength training volumes by means of the advanced computational modelling, biomechanical analysis and mobile monitoring technology. Of particular interest is the prediction of 1RM and the prediction of the ratio between hamstrings and quadriceps strength (H:Q ratio) compared against isokinetic strength tests as gold standard. Research has clearly shown that the quantification of 1RM is fundamentally important when it comes to the design of safe and efficient resistance training programs.

Secondary Objective: Assessment of changes in muscle size in the lower limbs due to different strength training volumes using the HMF technique. Of particular interest is the prediction of muscle volume using the HMF technique compared against data from MRI as gold standard, as well as the prediction of adaptation in hamstrings and quadriceps CSA due to the strength training intervention using HMF versus data from ultrasound, respectively.

Key baseline factors that will likely influence the primary and secondary endpoints are strength training experience and gender. The sample size and population group are specified to allow the analysis of gender-specific differences on study results. Thereby, the inclusion/exclusion criteria and study protocol, including a training-related questionnaire, are defined to minimize the bias of training experience.

Project design This project in sports science is designed as a confirmatory qualitative study in applied research involving healthy participants. The rationale of this project is to predict changes in muscle strength and muscle size due to strength training using computational modelling and mobile monitoring technology. In particular, the investigators will advance novel approaches in subject-specific anatomically-based modelling and mobile monitoring, which have previously tested in the research setting, and are now being applied to an intervention study in healthy volunteers to predict adaptations in muscle strength and muscle size in relation to strength training volume.

Study design: The specifics of the strength training intervention are carefully designed based on the current state of research in the field, and in line with strength training recommendations in musculoskeletal health, fitness and rehabilitation. In particular, the investigators will conduct an 8-week strength training intervention program of the key muscle-tendon groups associated with knee joint stability (hamstrings, quadriceps and triceps surae), with the study group (n=36, with 18F and 18M) being randomly allocated to different levels of training volume (Group#1: no training, Group#2: 1 training per week, Group#3: 3 trainings per week) with the same number of subjects and gender distribution in each group. Each participant will perform the strength training self-directedly in their chosen training-specific setting. Clear guidelines for warm-up, type and conduct of exercises will be given to all participants. The strength exercises are standard exercises for strengthening knee extension and flexion: squats, leg press, back extensions, heel raises, and single joint exercises.

Study parameters: Anthropometric parameters include body height, body weight, segmental circumferences, somatotype, body shape, muscle CSA and muscle volume of the lower limbs. Anthropometric parameters will be assessed by means of HMF fitting in combination with data from 3D body scanning and anthropometric measurements according to ISAK standards. Changes in CSA of the hamstrings and quadriceps will be compared between HMF and data from ultrasound before and after strength training intervention. Strength- and training-specific parameters include joint motion, joint acceleration, total joint moments, repetition count, 1RM and H:Q ratio. Strength- and training-specific parameters will be assessed by means of biomechanical analysis using data from optical motion capture and the iOS Strength Control app, and compared against data from isokinetic strength tests as gold standard. Additionally, data from MRI of the lower limbs will be acquired in a sub-group of 12 participants (6F, 6M).

PROJECT POPULATION AND STUDY PROCEDURES

Project population: The project population are healthy adult subjects who are all participating in their own strength training program on a regular weekly basis. The primary objective is to predict changes in muscle strength (i.e. primary outcome parameters: 1RM and H:Q ratio) following different training volumes of key muscle groups associated with knee joint stability. A power analysis was conducted using statistikguru.de to assess the required sample size for the primary outcome parameter, 1RM. Based on the power analysis, the investigators aim for a total of n=36 complete data sets (n=12 per study group of the strength training intervention), with a sub-group of n=12 participants additionally scheduled for MRI of the lower limbs at baseline.

The MRI-based assessment of muscle volume for validation of the HMF technique is analyzed independently from the strength training intervention. Thereby, the accuracy of the HMF technique is dependent on the initial generic musculoskeletal model that is used for model fitting, as well as the available subject-specific skin surface and anthropometric data.

All participants have to confirm their voluntary participation with a written informed consent before being submitted to any study procedure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants; and
* Age 20-40 years old; and
* No acute or chronic musculoskeletal symptoms or pain; and
* Experience with strength training (at least 1-year strength training experience with one training session per week or more); and
* Familiar with strength exercises of key muscles associated with knee joint stability.

Exclusion Criteria:

* Acute or chronic musculoskeletal pain; and/or
* Musculoskeletal surgery within the last 12 months; and/or
* Ongoing rehabilitation or treatment of musculoskeletal complaints or injury; and/or
* Neuromusculoskeletal disease (e.g. cerebral palsy); and/or
* Pregnancy.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in muscle strength in the lower limbs | 8 weeks
  one repetition maximum (1RM)
Changes in muscle strength in the lower limbs | 8 weeks
  Ratio hamstring to quadriceps force (H:Q ratio)

SECONDARY OUTCOMES:
Changes in muscle size of the lower limbs | 8 weeks
  Muscle volume
Changes in muscle size of the lower limbs | 8 weeks
  Muscle cross section area (CSA)

CONTACTS AND LOCATIONS:
Overall Officials: Silvio Lorenzetti, PD Dr., Principal Investigator — Swiss Federal Institute of Sport SFISM
Locations (1):
- Silvio Lorenzetti, Magglingen, Switzerland

IPD SHARING:
Plan to Share IPD: No